CLINICAL TRIAL: NCT06455917
Title: A Phase II Trial of Adoptive Cell Therapy With Tumor-infiltrating Lymphocytes in Patients With Non-Small Cell Lung Cancer
Brief Title: TIL Therapy in Non-small-cell Lung Cancer (NSCLC) Patients
Acronym: BaseTIL-02L
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-00254; th22Laeubli
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer; Lung Cancer (NSCLC)
Keywords: tumor-infiltrating lymphocytes; adoptive cell therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor-infiltrating lymphocyte product (TIL) transfer (Experimental): Tumor-specific T cells are expanded from excised tumor samples and stimulated in cell culture with interleukin-2 (IL-2). The resulting autologous TILs are then re-infused to the patient after a non-myeloablative lymphodepleting chemotherapy with cyclophosphamide and fludarabine. Activation of TILs in the patient is then supported by IL-2 administration. The transplant product will be produced in the Good Manufacturing Practice (GMP) facility of the University Hospital in Basel.
  Interventions: Drug: TILs（Tumor Infiltrating Lymphocytes）

INTERVENTIONS:
Drug: TILs（Tumor Infiltrating Lymphocytes） — The study procedures are:
  * Tumor collection: Study-specific intervention (eg, surgical resection and/or biopsy) to collect tumor material from one or more tumor lesions/metastases for the generation of the TIL product (tumor-infiltrating lymphocytes, TILs).
  * TIL expansion: Production of the TIL product in the Good-Manufacturing-Practice (GMP) Facility for Advanced Therapies of the University Hospital of Basel.
  * Lymphodepleting chemotherapy (lymphodepletion): Chemotherapy with cyclophosphamide and fludarabine (day -7 until day -3).
  * TIL transfer: Infusion of the TIL product back to the patient. TIL transfer is scheduled on day 0.
  * Interleukin-2 (IL-2) therapy: Therapy with high-dose IL-2 (Aldesleukin) every 8 hours for up to 15 doses. IL-2 therapy starts on day 0.

SUMMARY:
Aim of the study is to investigate the efficacy and safety of adoptive cell therapy (ACT) with tumor-infiltrating lymphocytes (TIL) in patients with advanced pre-treated non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Adoptive cell therapy (ACT) with tumor-infiltrating lymphocytes (TIL) is a personalized immunotherapy. TIL-ACT involves the infusion of autologous CD4+ and CD8+ T lymphocytes collected from tumor material and expanded ex-vivo with IL-2. These polyclonal immune cells can recognize and target multiple individualized tumor-specific antigens.

Clinical trials have demonstrated significant response rates in advanced melanoma patients. However, few trials have investigated TIL-ACT in other solid tumors, including NSCLC. For NSCLC patients experiencing disease progression after standard therapies (immune checkpoint inhibitors, targeted therapies), effective options are limited, often restricted to traditional chemotherapy with modest response rates, short durability, and significant toxicity. TIL-ACT represents an attractive individualized treatment approach for NSCLC patients.

The BaseTIL-02L study is a single-arm phase II trial investigating TIL-ACT efficacy in pretreated NSCLC patients. The study protocol includes preconditioning non-myeloablative chemotherapy (cyclophosphamide and fludarabine) and in-vivo TIL activation with high-dose interleukin 2 (for up to 15 doses, every 8 hours) following TIL transfer.

ELIGIBILITY:
Inclusion Criteria:

1. Ability of the patient to understand the purpose of the study, provide signed and dated informed consent prior to performing any protocol-related procedures (including screening evaluations), and be able and willing to comply with the study procedures.
2. Age ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1 (cf. Appendix).
4. Histologically confirmed NSCLC.
5. Disease progression after at least one standard therapy and without any approved curative-intended treatment option.
6. Accessible tumor lesion/metastasis for tumor collection.
7. Willingness of the patient to undergo a surgical intervention (eg, surgical resection and/or biopsy) to collect one or more tumor lesions/metastases.
8. Adequate organ function (pulmonary, cardiovascular, hematological, hepatic, and renal function) per investigator's judgment. Cardiac stress testing is required for all patients with underlying cardiac conditions and patients with age ≥ 50 years.
9. Negative serum pregnancy test in women of childbearing potential, in peri-menopausal women and in women with less than 2 years of menopause.

Exclusion Criteria:

1. Active central nervous system (CNS) metastases. Patients with stable CNS metastases ≥ 1 month after definitive treatment (eg, surgery and/or radiotherapy) are eligible.
2. Participants with an active second malignancy.
3. Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol, including autoimmune or immunodeficient conditions, significant pulmonary disease, significant cardiac and/or vascular disease per investigator's judgment.
4. Prior immune-related adverse events that would preclude re-challenge with an immune checkpoint inhibitor or immunomodulatory agent per investigator's judgment.
5. Immunosuppressive treatment that would preclude the patient from any of the study therapies per investigator's judgment.
6. Severe active infections or uncontrolled infectious conditions requiring treatment.
7. Any other conditions/diseases, allergies, dysfunctions, and/or findings, that would contraindicate the use of any of the study interventions or therapies.
8. Contraindication for any of the planned measures, interventions and/or treatments.
9. Pregnant or breastfeeding women, or female subject who are not willing to use an acceptable, highly effective method of contraception until the End-of-Study visit.
10. Known hypersensitivity to any of study therapies or drugs used for TIL production.
11. Known human immunodeficiency virus (HIV) infection (or tests positive for HIV 1 or 2 at Screening).
12. Known hepatitis B or hepatitis C infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free rate at 6 months after Tumor-infiltrating lymphocytes transfer. | 5-7 months after TIL transfer
  Progression-free rate (PFR) (RECIST v1.1 / iRECIST) at 6 months after TIL transfer, defined by the Kaplan-Meier estimator for progression-free survival (RECIST v1.1 / iRECIST) at 6 months (+/- 4 weeks as we allow this interval in the tumor assessment at 6 months).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to one year after TIL transfer
  The progression-free survival (PFS) is defined as the time from registration to objective tumor progression (determined by local investigators), or death due to any cause, whichever occurred first. PFS time for patients who have not progressed or died will be censored at the time of the last tumor assessment
Overall survival (OS) | up to one year after TIL transfer
  OS is defined as the time from registration to the date of death due to any cause
Severity of adverse events (CTCAE v5.0 criteria) | up to one year after TIL transfer
  Severity of adverse events (CTCAE v5.0 criteria) will be recorded to assess safety of combination of Tumor-infiltrating lymphocytes with IL-2
  CTCAE (Common Terminology Criteria for Adverse Events): Grade 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = fatal.
Objective response rate (ORR) | up to one year after TIL transfer
  ORR is defined as the proportion of patients with a best overall response of partial response or better (assessed by the local investigators
Duration of response (DOR) | up to one year after TIL transfer
  DOR is defined as the time from the first documented response and the date of the first documented tumor progression, death, or the last tumor assessment that occurred before subsequent therapy. DOR time for responders who have not progressed or died will be censored at the time of last tumor assessment
Frequency of adverse events (number) | up to one year after TIL transfer
  Frequency of adverse events (number) will be recorded to assess safety of combination of Tumor-infiltrating lymphocytes with IL-2
Incidence of adverse events (%) | up to one year after TIL transfer
  Incidence of adverse events (%) will be recorded to assess safety of combination of Tumor-infiltrating lymphocytes with IL-2

CONTACTS AND LOCATIONS:
Overall Officials: David König, Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Department of Medical Oncology, University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No